CLINICAL TRIAL: NCT02534506
Title: A Phase 1 Study of the Safety, Tolerability, Pharmacokinetics and Immunoregulatory Activity of Urelumab (BMS-663513) in Subjects With Advanced and/or Metastatic Malignant Tumors
Brief Title: Study of Urelumab in Subjects With Advanced and/or Metastatic Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA186-110
Record Dates: First submitted 2015-08-05; First posted 2015-08-27 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Malignant Tumors
Keywords: Advanced malignant tumors; Metastatic malignant tumors
MeSH Terms: conditions — Neoplasms | interventions — urelumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Urelumab (+ Nivolumab) intravenous (IV) infusion (Experimental)
  Interventions: Drug: Urelumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Urelumab
Drug: Nivolumab

SUMMARY:
The purpose of this study is to assess the safety and tolerability of BMS-663513 in subjects with advanced and/or metastatic malignant tumors.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects with previously treated advanced malignant solid tumor
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* For certain subjects, willing and able to provide pre-treatment tumor sample

Exclusion Criteria:

* Known or suspected central nervous system metastases or central nervous system as the only source of disease
* Other concomitant malignancies (with some exceptions per protocol)
* Active, known or suspected autoimmune disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2015-11-06 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-11 (Actual)

PRIMARY OUTCOMES:
Safety of urelumab monotherapy as measured by the dose limiting toxicity (DLT) in subjects with advanced and/or metastatic malignant tumors | From day 1 of treatment up to 60 days of follow-up
Safety of urelumab monotherapy as measured by adverse events (AEs) and serious adverse events (SAEs) in subjects with advanced and/or metastatic malignant tumors | From day 1 of treatment up to 60 days of follow-up
Tolerability of urelumab monotherapy as measured by the DLT in subjects with advanced and/or metastatic malignant tumors | From day 1 of treatment up to 60 days of follow-up
Tolerability of urelumab monotherapy as measured by AEs and SAEs in subjects with advanced and/or metastatic malignant tumors | From day 1 of treatment up to 60 days of follow-up

SECONDARY OUTCOMES:
Safety of urelumab-nivolumab combination therapy as measured by AEs and SAEs in subjects with advanced and/or metastatic malignant tumors | From day 1 of treatment up to 100 days of follow-up
Tolerability of urelumab-nivolumab combination therapy as measured by AEs and SAEs in subjects with advanced and/or metastatic malignant tumors | From day 1 of treatment up to 100 days of follow-up
Cmax (Maximum observed serum concentration) of urelumab when administered alone | Cycle 1, 2, 3, 4, 5, 6, 7, 12, 16, up to 60 days of follow up
  21 days/cycle for Urelumab monotherapy
Ctrough (Trough observed serum concentration) of urelumab when administered alone | Cycle 1, 2, 3, 4, 5, 6, 7, 12, 16, up to 60 days of follow up
  21 days/cycle for Urelumab monotherapy
Tmax (Time of maximum observed serum concentration) of urelumab when administered alone | Cycle 1, 2, 3, 4, 5, 6, 7, 12, 16, up to 60 days of follow up
  21 days/cycle for Urelumab monotherapy
AUC(0-T) [Area under the concentration-time curve from time zero to the last quantifiable concentration] of urelumab when administered alone | Cycle 1, 2, 3, 4, 5, 6, 7, 12, 16, up to 60 days of follow up
  21 days/cycle for Urelumab monotherapy
AUC(TAU) [Area under the concentration-time curve in one dosing interval] of urelumab when administered alone | Cycle 1, 2, 3, 4, 5, 6, 7, 12, 16, up to 60 days of follow up
  21 days/cycle for Urelumab monotherapy
AUC(INF) [Area under the concentration-time curve from time zero to infinity and the extrapolated area] of urelumab when administered alone | Cycle 1, 2, 3, 4, 5, 6, 7, 12, 16, up to 60 days of follow up
  21 days/cycle for Urelumab monotherapy
T-HALF (Elimination half life) of urelumab when administered alone | Cycle 1, 2, 3, 4, 5, 6, 7, 12, 16, up to 60 days of follow up
  21 days/cycle for Urelumab monotherapy
CLT (Total body clearance) of urelumab when administered alone | Cycle 1, 2, 3, 4, 5, 6, 7, 12, 16, up to 60 days of follow up
  21 days/cycle for Urelumab monotherapy
Vss (Volume of distribution at steady state) of urelumab when administered alone | Cycle 1, 2, 3, 4, 5, 6, 7, 12, 16, up to 60 days of follow up
  21 days/cycle for Urelumab monotherapy
AI (Accumulation Index: ratio of AUC(TAU) and Cmax in cycle at steady state to those after the first cycle) of urelumab when administered alone | Cycle 1, 2, 3, 4, 5, 6, 7, 12, 16, up to 60 days of follow up
  21 days/cycle for Urelumab monotherapy
Cmax of urelumab when co-administered | Cycle 1, 2, 3, 4, 5, 6, 9, up to 100 days of follow up
  28 days/cycle for combination therapy of Urelumab and Nivolumab
Coeff of urelumab when co-administered | Cycle 1, 2, 3, 4, 5, 6, 9, up to 100 days of follow up
  28 days/cycle for combination therapy of Urelumab and Nivolumab
Ctrough of urelumab and nivolumab when co-administered | Cycle 1, 2, 3, 4, 5, 6, 9, up to 100 days of follow up
  28 days/cycle for combination therapy of Urelumab and Nivolumab
Tmax of urelumab and nivolumab when co-administered | Cycle 1, 2, 3, 4, 5, 6, 9, up to 100 days of follow up
  28 days/cycle for combination therapy of Urelumab and Nivolumab
AUC(0-T) of urelumab and nivolumab when co-administered | Cycle 1, 2, 3, 4, 5, 6, 9, up to 100 days of follow up
  28 days/cycle for combination therapy of Urelumab and Nivolumab
AUC(TAU) of urelumab and nivolumab when co-administered | Cycle 1, 2, 3, 4, 5, 6, 9, up to 100 days of follow up
  28 days/cycle for combination therapy of Urelumab and Nivolumab
AUC(INF) of urelumab and nivolumab when co-administered | Cycle 1, 2, 3, 4, 5, 6, 9, up to 100 days of follow up
  28 days/cycle for combination therapy of Urelumab and Nivolumab
T-HALF of urelumab when co-administered | Cycle 1, 2, 3, 4, 5, 6, 9, up to 100 days of follow up
  28 days/cycle for combination therapy of Urelumab and Nivolumab
CLT of urelumab when co-administered | Cycle 1, 2, 3, 4, 5, 6, 9, up to 100 days of follow up
  28 days/cycle for combination therapy of Urelumab and Nivolumab
Vss of urelumab when co-administered | Cycle 1, 2, 3, 4, 5, 6, 9, up to 100 days of follow up
  28 days/cycle for combination therapy of Urelumab and Nivolumab
Anti-drug Antibody (ADA) status of the subject in response to Urelumab when administered alone | Cycle 1, 2, 4, 8, 12, 16, up to 60 days of follow up
  21 days/cycle for Urelumab monotherapy
ADA status of the subject in response to Urelumab and Nivolumab when co-administered | Cycle 1, 2, 4, 5, 9, up to 100 days of follow up
  28 days/cycle for combination therapy of Urelumab and Nivolumab
Best overall response (BOR) of urelumab monotherapy | Every 6-8 weeks during the treatment period
BOR of urelumab and nivolumab combination therapy | Every 6-8 weeks during the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Kobe, Hyōgo, Japan

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx